CLINICAL TRIAL: NCT00594932
Title: Biomarker-Linked Outcomes of Cellcept in Lupus Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oklahoma Medical Research Foundation (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMRF 06-23; Aspreva Pharmaceuticals grant (Other Grant/Funding Number: Aspreva Pharmaceutical Investigator-Initiated Study)
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Systemic Lupus Erythematosus; Arthritis
Keywords: lupus, arthritis, mycophenolate, biomarkers
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: (Active Comparator): Participants randomly assigned to Arm I will receive mycophenolate mofetil in ascending doses during Month 1, and 3 grams/day (or less if there are tolerance issues) for Months 2 through 6. During Month 1 these participants receive the same number of pills as every other month, but with ascending doses of mycophenolate mofetil and descending numbers of placebo pills. Week one for a total of 1.5 gm/day of mycophenolate mofetil, Week two 2.0 gm/day, Week three 2.5 gm/day and Week 4 3 gm/day. Dose can be held or decreased for tolerance issues at any time.
  Interventions: Drug: mycophenolate mofetil
- Arm 2 (Placebo Comparator): Patients Randomly Assigned to Arm 2 will receive a placebo comparator. The placebo treatment will be structured so that they will undergo the same type of dosing in Month 1 that the ascending dose patient from Arm 1 undergo, but will have placebo in both bottles of pills. At the end of three months, after assessment of primary outcome, these patients enter open label treatment for three more months. During the fourth month this group continues to receive the same number of pills as they received before, with ascending doses of mycophenolate mofetil given vs descending placebo pills so that their induction is the same as those in Arm 1 at the first month.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: mycophenolate mofetil — First treatment month: mycophenolate mofetil ascending doses orally Second treatment month to end of study: mycophenolate mofetil 3 gms/day (or less if tolerance issues arise)
  Other Names: mycophenolate; Cellcept
  Arms: Arm I:
Other: placebo — oral placebo will be given in ascending "doses" during the first month and at full "dose" during the second and third month (or at lower "dose" if tolerance issues warrant). During the fourth month mycophenolate mofetil will be given in ascending doses to 3 gms/day (or less if tolerance issues arise) and continues until the end of the study at 6 months.
  Other Names: inert tablet; oral placebo pill
  Arms: Arm 2

SUMMARY:
We hypothesize that mycophenolate mofetil(Cellcept)is safe and effective for lupus arthritis. In this study, patients with lupus will be randomly assigned to receive mycophenolate mofetil or placebo (inert pills) for three months. At the end of three months all patients will receive mycophenolate mofetil for three additional months. The effectiveness on arthritis and other symptoms of lupus will be measured by joint counts and by the BILAG instrument (a measure of overall lupus disease activity. Additionally special blood tests aimed at understanding the biologic effects of mycophenolate mofetil will also be performed at some visits. The primary outcome measurement will be the safety and effectiveness of this treatment (as compared to placebo) at the three month point. The trial will continue in a blinded fashion (neither the investigator or the participants know who is getting mycophenolate and who is getting placebo) until 24 patients have completed the first three months of the protocol.

DETAILED DESCRIPTION:
Patients and Methods:

27 patients with active BILAG B or A arthritis, with at least 6 swollen and 6 tender joints entered a six month study of MMF vs placebo for three months followed by open label MMF. 14 patients (12 women and 2 men) received placebo at baseline and 13 patients (11 women and 2 men) received MMF. Primary Outcome was Major Clinical Response at 3 months, then all patients received open label Cellcept for another 3 months. Blood was drawn for safety, lupus disease activity measures and exploratory Biomarkers, Joint counts were performed monthly. At baseline background DMARDs were stopped. Plaquenil was allowed. All patients received 160 mg depomedrol at baseline and were allowed 80 mg shots at subsequent months after blood draws and procedures had been completed.

DEFINITION of RESPONSE

Prespecified Primary Endpoint: Complete Clinical Response:

BILAG C in musculoskeletal by Week 12 and decrease to 0.25 or less of tender +swollen jt counts

Prespecified Secondary Endpoint: Partial response:

One letter drop in musculoskeletal by Week 12 OR decrease to 0.5 or less tender + swollen jt counts

Exploratory Measure (not prespecified): Major Clinical Response:

BILAG C in musculoskeletal by Week 12 and decrease to 0.5 or less of tender +swollen jt counts. (In the primary analysis the one patient who met this endpoint was designated as a partial responder since those prespecified criteria were also met.

Non response:

Does not meet above criteria for complete or partial response

Additional Measures: (prespecified secondary endpoints) included joint counts, changes in BILAG and SLEDAI and physician and patient global assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SLE by the 1995 modification of revised ACR criteria (includes antiphospholipid antibodies)
2. BILAG A arthritis or BILAG B arthritis with at least 6 tender and 4 swollen joints at screening and baseline
3. Stable prednisone dose at 20 mg of less for one month at baseline.
4. If on antimalarials must be stable for at least one month at baseline
5. If on NSAIDS must be on a stable regimen for at least one month but can be prn dosing
6. Must be willing to withdraw from azathioprine or MTX at the time of screening.
7. Between ages 14 and 70
8. Women of childbearing potential must have a negative pregnancy test at screening and at each month during the study.
9. All participants (male and female) must, if fertile, agree to practice contraception during the entire course of the study. This may include barrier, oral contraceptives, depo-provera, intrauterine device and/or abstinence.

   -

Exclusion Criteria:

1. Inability to understand informed consent
2. Drug or alcohol abuse within the past six months
3. In the opinion of the investigator, it is not likely the patient can comply with the protocol for any reason, or participation in the protocol is not in the patient's best interest.
4. Unstable medical condition that, in the opinion of the investigator would contraindicate study participation
5. History of malignancy (except for basal cell carcinoma at any time and/or cervical cancer or squamous cell cancer at least five years previous to screening).
6. Use of cyclosporine, leflunomide, cyclophosphamide or ay biologic agent within three months prior to screening.
7. Participation in any clinical study of an investigational agent within three months of screening -

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan T. Merrill, M.D., Principal Investigator — Oklahoma Medical Research Foundation; Robert Clancy, PhD, Study Chair — NYU Langone Health
Locations (1):
- Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 patients with SLE and active arthritis (with or without other manifestations) were randomized 1:1 to receive mycophenolate mofetil (MMF) or placebo. A total of 13 received MMF and 14 received placebo for the first 3 months. For the second three months patients could elect to continue on open lable MMF
Pre-assignment Details: Patients were excluded if they did not have arthritis sufficient to be treated with an aggressive immune suppressant. All patients were offered steroid rescue at baseline, those who required immediate treatment and/or who could not be given steroids were excluded from the study
Groups:
- Patients Who Received MMF for the First 3 Months: 13 patients were randomized to receive MMF for the first 3 months. MMF was (blindly) increased to maximal tolerated dose or 3 gms/daily whichever was lowest.
- Patients Who Received Placebo for the First 3 Months: 14 patients were randomized to placebo for the first three months
Period: First 3 Months
Arm/Group | Patients Who Received MMF for the First 3 Months | Patients Who Received Placebo for the First 3 Months
Started | 13 | 14
Completed | 12 | 11
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3
Period: Final 3 Months
Arm/Group | Patients Who Received MMF for the First 3 Months | Patients Who Received Placebo for the First 3 Months
Started | 12 | 11
Completed | 8 | 8
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Who Received MMF for the First 3 Months | Patients Who Received Placebo for the First 3 Months | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (9.42) | 34.0 (11.35) | 36.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Arthritis Complete Response
Description: Complete response at three months (This is defined as </= 0.25 of the total tender plus swollen joints observed at baseline and British Isles Lupus Assessment Group (BILAG) index C (mild) or D (no longer present) score in the Musculoskeletal system), comparing treatment to placebo group as complete responder or not complete responder. This was an intent to treat analysis so dropouts were counted as non-responders.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Patients Who Received MMF for the First 3 Months | Patients Who Received Placebo for the First 3 Months
Number analyzed (Participants) | 13 | 14
participants | 4 | 0

2. Secondary Outcome: Major Arthritis Response
Description: This is defined as at least a 50% reduction in tender + swollen joint counts and severity rated as mild as defined by the British Isles Lupus Assessment Group Index
Time Frame: 3 months
Population: All those randomized to MMF or placebo
Measure: Number; unit: participants
Arm/Group | Patients Who Received MMF for the First 3 Months | Patients Who Received Placebo for the First 3 Months
Number analyzed (Participants) | 13 | 14
participants | 5 | 0
Statistical Analysis 1: Comparison: Patients Who Received MMF for the First 3 Months vs Patients Who Received Placebo for the First 3 Months; this is a categorical assessment. Prespecified. Fishers exact test. Significant is calculated as < 0.05; Test type: Superiority or Other; p = 0.041, Fisher Exact — This was the primary endpoint therefore no adjustment for multiple comparisons was necessary; superiority = 4

3. Secondary Outcome: Major and Partial Clinical Response
Description: Those meeting the Criteria for Major or Complete Clinical Response as listed in the preceding endpoints or who meet criteria for partial response defined as at least a 25% decrease in tender and swollen joint count and improvement of at least one severity rating for arthritis as at least one level on the British Isles Lupus Assessment Group Index.
Time Frame: 3 Months
Population: Patients who entered and were randomized to receive MMF vs Placebo.
Measure: Number; unit: participants
Arm/Group | Patients Who Received MMF for the First 3 Months | Patients Who Received Placebo for the First 3 Months
Number analyzed (Participants) | 13 | 14
participants | 9 | 5

ADVERSE EVENTS:
Time Frame: 3 months for non serious adverse events and six months for deaths and serious adverse events. We did not formally collect adverse events after the end of the double blind part of the study since all continuing patients received open lable MMF, a standard of care for SLE. Since we are confident that there were no additional deaths or serious adverse events over six months, we can report those for the entire six month period but we only have non serious adverse events collected for three months.
Description: Definitions do not differ. However we only collected accurate non-serious adverse events for the first three months. After that it was no longer a blinded trial, those who wanted to continue were receiving MMF, a standard of care for SLE. Safety of this commonly used drug would not be interpretable in a tiny trial after the double blind period. However, we can report SAEs for six months, since we are confident we can be accurate about those. There were also no deaths over six months.
Groups:
- Mycophenolate Mofetil: Patients receiving mycophenolate mofetil from baseline throughout their participation in the study (up to six months). Mycophenolate is a standard of care treatment for SLE, and the primary endpoint was at three months, after which mycophenolate was given "open lable." This trial did not collect adverse events after three months in any formal manner that can be reported here.
  However there were no deaths so we can report that for six months. We can also report serious adverse events for all six months. Therefore deaths and serious adverse events are reported for six months and placebo crossovers are included in the "at risk" population for a total of 24 at risk. However non serious adverse events can only be reported for three months so the population at risk remains at 13 for non serious adverse events.
- Placebo: Patients receiving placebo for the first three months. They were then offered mycophenolate mofetil for up to three more months. Since this is a standard of care for SLE formal assessment of adverse events was not performed during the second three months. We cannot provide any data after the first three months on placebo patients since there were no placebo patients after the first three months. Therefore the at risk population on placebo is 14 and the reporting period is 3 months for them. This is true for all types of adverse events since there was no placebo group after 3 months.
Arm/Group | Mycophenolate Mofetil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/14
Serious Adverse Events (participants affected / at risk) | 2/24 | 2/14
Other Adverse Events (participants affected / at risk) | 12/13 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (N=24) | Placebo (N=14)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient hospitalized but cardiac cause of chest pain ruled out
upper GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) — one patient in the MMF treated group had an upper GI bleed and the condition resolved with supportive care
groin abcess (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Groin abcess in a placebo patient
avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — avascular necrosis in a placebo patient
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (N=13) | Placebo (N=14)
mild to moderate infection (includes respiratory tract, urinary tract, vaginitis, non serious abcess (Infections and infestations) | 9 (16) | 8 (13)
gastroenteritis (Gastrointestinal disorders) | 8 (15) | 5 (9)
Other mild or moderate AEs (General disorders) | 7 (7) | 12 (13)
Renal Stones (Metabolism and nutrition disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No